CLINICAL TRIAL: NCT00681902
Title: Jet Lidocaine for Pain Relief During Needle Insertion in a Pediatric Emergency Department.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Marc Auerbach, Fellow Pediatric Emergency Medicine, Department of Pediatrics, NYUSOM
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-705
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Pain
Keywords: Pediatric; Pain; Needle; Emergency; Phlebotomy; Intravenous; Lidocaine; Local; Anesthesia
MeSH Terms: conditions — Pain; Emergencies | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Jet lidocaine
  Interventions: Drug: Lidocaine
- 2 (Placebo Comparator): Jet saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Jet lidocaine compared to jet placebo before needle insertion
  Other Names: National medical jet injector system
  Arms: 1
Drug: Placebo — Jet saline
  Arms: 2

SUMMARY:
The purpose of this study is to explore to what degree, if any, Jet lidocaine will reduce or alleviate pain, as compared to Jet normal saline, in children undergoing needle insertion in the Pediatric Emergency Department (PED). If effective, Jet lidocaine would afford a novel rapidly acting local anesthesic for children in the PED.

DETAILED DESCRIPTION:
This randomized clinical trial involves double blind allocation of either (1) Jet administration of buffered 1% lidocaine or (2) Jet normal saline (placebo) prior to needle insertion in the PED. The product will be prepackaged on a weekly basis at an off site pharmacy into the jet injector system and all devices will be labeled as "study drug" with an assigned number. We estimate 30 patients being enrolled in each one-month period and the pharmacy will allocate 10 devices of study medication and 10 devices of normal saline. Our estimated sample size is 84 patients per group. The study duration will continue until the sample size is achieved. An interim analysis of data will be performed after 25% or 21 patients are obtained in each group.

A total of 168 patients will be expected to participate in order to achieve our sample size. The a priori sample size analysis uses a two tailed student's t-test with an alpha of 0.05 and a power of The study is open to children of any race or ethnicity. There will be no race or ethnicity-based enrollment restrictions or selection factors for the population to be included in this study.

All children presenting to the Pediatric Emergency Department at Bellevue Hospital are first triaged by the nursing staff. Triage includes documenting vital signs, a chief complaint, and a brief clinical assessment. The physician (resident, fellow, or attending) evaluates the patient and repeats a more extensive clinical assessment. Children with clinical evaluations and treatment plans that identify a need for needle insertion will be prepared for the procedure by a physician, nurse, and/or a Certified Child Life Specialist (CCLS). Preparation involves education and support to the parent and/or child before and during the procedure. The pre-procedure preparation is a part of the routine care for all children who present to the PED and require a procedural intervention.

Patients will be randomly assigned to receive one of two treatments prior to the procedure. The treatment group will receive 0.2 cc of 1% buffered lidocaine via Jet injection, while the control group will receive 0.2 cc of normal saline via Jet injection. All patients who fulfill enrollment criteria and with whom consent and assent (if appropriate) are obtained will be assigned consecutively.

1. The provider's decision to insert a needle is determined as part of the patient's standard care for the diagnosis or treatment of illness. A standard history and physical examination will be performed by the ED physician/nurse and includes information sufficient to determine patient eligibility. All children undergoing needle insertion will be assessed for eligibility by a trained provider based on information routinely documented (see above Inclusion/Exclusion Criteria). Children eligible to receive EMLA cream will be excluded and will receive EMLA cream routinely. Other anesthetics or analgesics will not be withheld from any patient enrolled in this study. The standard pre-procedure preparation time will provide an appropriate time period to educate the patient and parent about the study and obtain consent. This process will not delay the patient's care. Standard non-pharmacologic emotional support and explanations will be provided to the patient and/or parent.
2. For patients meeting inclusion criteria, informed consent will be obtained from the parent or legal guardian. Patients who are 18 years of age will provide their own consent. Informed assent will also be obtained in children less than 18 years of age. Consent and assent will be obtained during the standard pre-procedural preparation time.
3. If informed consent/assent is obtained, the patient and parent will receive additional education about the Jet device. This patient will undergo standard needle insertion by a trained provider and concomitantly receive supportive care including, but not limited to, age appropriate education, distraction, relaxation, and support.
4. A Color Analogue pain score (CAS) (see outcome measures section for CAS background and description, and fig 2) will be obtained from the patient at the baseline, prior to the start of the procedure. The Jet application will occur at the insertion site, prior to the needle being inserted into the skin. A CAS pain score will be obtained from the patient subsequent to administration of the device. The provider will wait thirty seconds prior to insertion of the needle into the skin. A CAS pain score for needle insertion will be collected after completion of the procedure. After one minute a post procedure CAS score will be collected. The parent and/or support staff will be with the child throughout the entire procedure.
5. After the procedure the provider will document patient demographics, diagnosis, and Likert scales for cooperation and ease of insertion (see provider document). The provider will ask the parent and child one question related to satisfaction after the completion of the procedure.
6. Patients will be withdrawn from the study if either the patient or caregiver requests withdrawal at any time.
7. After insertion of the needle appropriate diagnostic and therapeutic interventions will be continued leading to either hospital admission with the IV or discharge home with removal of the IV upon discharge.

The J-Tip Jet device (National Medical Products, CA) will be purchased as an empty device and sent to Dr. Nayan Patel at Central Drugs Pharmacy, CA, for preparation. Central Drugs Pharmacy will fill these devices and ship them to Bellevue hospital. The devices will be filled and packaged, using aseptic techniques, with either 0.25 cc of normal saline or 0.25 cc of 1% buffered lidocaine. This device is FDA approved for administration of lidocaine in children and is currently used in a number of other institutions at the time of this study.

Pain, the primary outcome, will be assessed using the Color Analogue pain Scale (CAS) (1-5) (see appendix for CAS scale picture). This scale is anchored by descriptors "no pain" and "most pain" with gradation in color, area, and length (see attached CAS figure). The point on the tool that is identified by the child with the plastic marker on the colored scale front side is converted to a corresponding numerical scale from the back of the tool. This number is the CAS score in centimeters. This scale has been well validated for use in children over five years of age undergoing procedures in the PED with minimal or no training with this tool. The following instructions are given prior to use of the scale: "This is a pain scale. The bottom, where it is small and white, means no pain, and the top, where it is wider and red, means the most pain you can imagine (instructor points to anchor). You slide the marker to the spot on the scale that shows how much pain you are having right now. (2)"

The CAS pain scale will be self-reported by the patient at the site of needle insertion at a number of points in time. A 2.5 cm change in CAS is considered clinically significant (11).

1. Pre-Jet
2. Jet administration
3. Insertion of needle into the skin (60 seconds after Jet)
4. Post-needle insertion (1 minutes after completion of insertion)

Secondary outcomes will be measured to assess satisfaction. All patients and parents will be asked "Based on your IV start today, would you like this numbing medicine in the future?" (8) The provider will report satisfaction related to cooperation and "difficulty of finding a vein" using a 5-point likert scales. The patient's demographic data, location of placement, diagnosis, and number of attempts will be included in the study documentation.

All data collection sheets will be filed in a locked collection cabinet, to be reviewed only by the principal investigators after completion. Study number and age will be identified on the data collection document.

Each child's data collection sheets (See Data Collection Forms) will include their gender, ethnicity, date of visit, age, pain scores, and survey data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 - 18 years
2. Evaluation and treatment requiring needle insertion in <60 minutes (Patient is not a candidate for EMLA cream)
3. Parent or patient consent, and child assent

Exclusion Criteria:

1. Age <5 years or >18 years
2. Children eligible for or receiving EMLA cream
3. Significant blunt or penetrating trauma requiring rapid evaluation/resuscitation (GCS<15)
4. Unstable shock
5. Altered sensorium or intoxication
6. History of allergy to Lidocaine
7. Neurologic deficit involving a lack of sensation in area of insertion
8. Developmental delay so as not to understand pain scale

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Pain, the primary outcome, will be assessed using the Color Analogue pain Scale before and after needle insertion in each group and compared for a clinically significant difference. | Primary outcome was measured at time of initial needlestick in ED

SECONDARY OUTCOMES:
Provider and patient satisfaction. | Secondary outcome was measured at time of initial needlestick in ED.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mojica, Principal Investigator — NYU/Bellevue
Locations (1):
- Bellevue Hospital, New York, New York, United States